CLINICAL TRIAL: NCT05915520
Title: Baduanjin Program Effect on Geriatric Functional Dyspepsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Internal Medicine and Geriatrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004557
Record Dates: First submitted 2023-06-13; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — Pantoprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): the 20-geriatric group will receive 5-session per-week 40-minute baduinjuin for 8 weeks plus the daily dose of pantoprazole (40 mg orally administered tablet drug)
  Interventions: Behavioral: baduinjuin activities
- group B (Other): this 20-geriatric group will receive the daily dose of pantoprazole (40 mg orally administered tablet drug for 8 weeks .
  Interventions: Other: pantoprazole

INTERVENTIONS:
Behavioral: baduinjuin activities — in this 20-geriatric group will receive 5-session per-week 40-minute baduinjuin for 8 weeks plus the daily dose of pantoprazole (40 mg orally administered tablet drug)
  Arms: group A
Other: pantoprazole — in this 20-geriatric group will receive the daily dose of pantoprazole (40 mg orally administered tablet drug for 8 weeks .
  Arms: group B

SUMMARY:
functional dyspepsia is very common between geriatric population

DETAILED DESCRIPTION:
Forty Egyptian geriatrics with functional dyspepsia, after randomization, will be divided to 2 groups; the first 20-geriatric group will receive 5-session per-week 40-minute baduinjuin for 8 weeks plus the daily dose of pantoprazole (40 mg orally administered tablet drug. in the other 20-geriatric group, the daily dose of drug will be administered only for 8 weeks .

ELIGIBILITY:
Inclusion Criteria:

* functional dyspepsia complaints
* geriatric population

Exclusion Criteria:

* cardiac complaints
* respiratory complaints
* articular complaints

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
cortisol | It will be measured after 8 weeks
  it is a serum stress marker

SECONDARY OUTCOMES:
depression sub component of Hospital anxiety and depression scale | It will be measured after 8 weeks
  It will be measure depression
anxiety sub component of Hospital anxiety and depression scale | It will be measured after 8 weeks
  It will be measure anxiety
Glasgow dyspepsia severity score | It will be measured after 8 weeks
  It will be used to assess functional dyspepsia
visual analogue scale | It will be measured after 8 weeks
  It will be used to assess abdominal symptoms of geriatric patients regarding functional dyspepsia

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt